CLINICAL TRIAL: NCT02630459
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of AMG 334 in Migraine Prevention
Brief Title: A Safety and Efficacy Study to Evaluate AMG 334 in Migraine Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20120309
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Migraine
Keywords: Migraine Prevention; Headache; Prophylaxis
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — erenumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Double Blind Treatment Phase (DBTP): Placebo (Placebo Comparator): Participants received placebo by subcutaneous injection on day 1 and at weeks 4, 8, 12, 16, and 20 in the double-blind treatment phase.
  Interventions: Drug: Placebo
- DBTP: Erenumab 28 mg QM (Experimental): Participants received erenumab 28 mg by subcutaneous injection on day 1 and at weeks 4, 8, 12, 16, and 20 in the double-blind treatment phase.
  Interventions: Drug: Erenumab
- DBTP: Erenumab 70 mg QM (Experimental): Participants received erenumab 70 mg by subcutaneous injection on day 1 and at weeks 4, 8, 12, 16, and 20 in the double-blind treatment phase.
  Interventions: Drug: Erenumab
- DBTP: Erenumab 140 mg QM (Experimental): Participants received erenumab 140 mg by subcutaneous injection on day 1 and at weeks 4, 8, 12, 16, and 20 in the double-blind treatment phase.
  Interventions: Drug: Erenumab
- Open-Label Treatment Phase (OLTP): Erenumab 70-140 mg QM (Experimental): Participants received an erenumab dose of 70 and/or 140 mg QM SC (depending on the participant's visit completion status after Institutional Review Board [IRB] approval of Protocol Amendment 2) in the OLTP for a total of 76 weeks.
  Interventions: Drug: Erenumab
- CHU Sub-Study: Two 70 mg/mL AI/pens (Experimental): A subset of participants in the OLTP randomized to self administer erenumab via two 70 mg/mL autoinjector (AI)/pens on day 29 and day 57 of the CHU Sub-Study
  Interventions: Drug: Erenumab
- CHU Sub-Study: One 140 mg/mL AI/pen (Experimental): A subset of participants in the OLTP randomized to self administer erenumab via one 140 mg/mL AI/pen on day 29 and day 57 of the CHU Sub-Study
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Placebo — placebo via subcutaneous injection
  Arms: Double Blind Treatment Phase (DBTP): Placebo
Drug: Erenumab — erenumab via subcutaneous injection
  Other Names: AMG 334, Aimovig™
  Arms: DBTP: Erenumab 140 mg QM; DBTP: Erenumab 28 mg QM; DBTP: Erenumab 70 mg QM; Open-Label Treatment Phase (OLTP): Erenumab 70-140 mg QM
Drug: Erenumab — erenumab via autoinjector (AI)/pen
  Other Names: AMG 334, Aimovig™
  Arms: CHU Sub-Study: One 140 mg/mL AI/pen; CHU Sub-Study: Two 70 mg/mL AI/pens

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel-group, multicenter study followed by an open-label treatment phase (OLTP). To evaluate the effect of erenumab (AMG 334) compared to placebo on the change from baseline in monthly migraine days.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled study in participants with episodic migraine. The study's double blind treatment phase (DBTP) is designed to evaluate if treatment with erenumab once a month for 6 months compared with placebo is effective in reducing the mean monthly migraine days. Additionally, this study will continue to evaluate the efficacy and safety of erenumab during the OLTP where participants will continue to receive active treatment monthly.

The study also includes a clinical home use (CHU) sub-study to assess a participant's ability to self-administer 140 mg of erenumab. Participants will be randomized 1:1 to use either 2 pre-filled 70 mg/mL autoinjector (AI)/pens or 1 pre-filled 140 mg/mL AI/pen. Participation in the substudy is optional, and no additional samples will be collected for the sub-study.

After implementation of Protocol Amendment 2, the dose of erenumab in the OLTP increased from 70 mg to 140 mg QM. Participants who had already completed week 48 remain on 70 mg QM, participants not yet starting the OLTP, or not yet completing the week 48 visit receive erenumab 140 mg QM for the remainder of the OLTP.

ELIGIBILITY:
Inclusion Criteria to be assessed prior to entering the subject into the initial screening and/or baseline phase:

* Provided informed consent prior to initiation of any study-specific activities/procedures
* History of migraine (with or without aura) for ≥ 12 months prior to screening according to the International Headache Society (IHS) Classification The International Classification of Headache Disorders (ICHD)-3 (Headache Classification Committee of the IHS, 2013),
* Migraine frequency: ≥ 4 and < 15 migraine days per month on average across the 3 months prior to screening,
* Headache frequency: < 15 headache days per month on average across the 3 months prior to screening.

Inclusion Criteria to be assessed during the baseline phase and confirmed prior to randomizing the subject into the double-blind treatment phase:

* Demonstrated at least 80% compliance with the electronic Diary (eDiary),
* Migraine frequency: ≥ 4 and < 15 migraine days during the baseline phase based on the eDiary calculations,
* Headache frequency: < 15 headache days during the baseline phase based on the eDiary calculations.

Inclusion Criteria for the Clinical Home Use (CHU) Substudy:

- Subjects must have provided informed consent for the substudy. Subjects enrolling in the CHU substudy must have received open-label 140 mg erenumab for at least 1 dose.

Exclusion Criteria:

* Older than 50 years of age at migraine onset,
* History of cluster headache or hemiplegic migraine headache,
* Unable to differentiate migraine from other headaches,
* No therapeutic response with > 2 of the following 7 medication categories for prophylactic treatment of migraine after an adequate therapeutic trial: Category 1: Divalproex sodium, sodium valproate, Category 2: Topiramate, Category 3: Beta blockers (for example: atenolol, bisoprolol, metoprolol, nadolol, nebivolol, pindolol, propranolol, timolol), Category 4: Tricyclic antidepressants (for example: amitriptyline, nortriptyline, protriptyline),Category 5: Serotonin-norepinephrine reuptake inhibitors (for example: venlafaxine, desvenlafaxine, duloxetine, milnacipran), Category 6: Flunarizine, verapamil, lomerizine, Category 7: Lisinopril, candesartan,
* Used a prohibited medication, device or procedure within 2 months prior to the start of the baseline phase or during the baseline phase,
* Received botulinum toxin in the head and/or neck region within 4 months prior to the start of the baseline phase or during the baseline phase,
* Taken the following for any indication in any month during the 2 months prior to the start of the baseline phase: Ergotamines or triptans on ≥ 10 days per month, or Simple analgesics (nonsteroidal anti-inflammatory drugs [NSAIDs], acetaminophen) on ≥ 15 days per month, or Opioid- or butalbital-containing analgesics on ≥ 4 days per month,
* Anticipated to require any excluded medication, device or procedure during the study,
* Active chronic pain syndromes (such as fibromyalgia and chronic pelvic pain),
* History of major psychiatric disorder (such as schizophrenia and bipolar disorder), or current evidence of depression based on a Beck Depression Inventory (BDI)-II total score > 19 at screening. Subjects with anxiety disorder and/or major depressive disorder are permitted in the study if they are considered by the investigator to be stable and are taking no more than 1 medication for each disorder. Subjects must have been on a stable dose within the 3 months prior to the start of the baseline phase,
* History of seizure disorder or other significant neurological conditions other than migraine. Note: A single childhood febrile seizure is not exclusionary,
* Malignancy within the 5 years prior to screening, except non melanoma skin cancers, cervical or breast ductal carcinoma in situ,
* Human immunodeficiency virus (HIV) infection by history,
* Hepatic disease by history, or total bilirubin (TBL) ≥ 2.0 x upper limit of normal (ULN) or alanine transaminase (ALT) or aspartate aminotransferase (AST) ≥ 3.0 x ULN, as assessed by the central laboratory at initial screening, or evidence of acute or chronic hepatitis B or hepatitis C virus. Hepatitis status will be evaluated by testing for hepatitis B surface antigen (HepBsAg), total hepatitis B core antibody (HepBcAb) and hepatitis C antibody by the central laboratory at initial screening. Polymerase chain reaction (PCR) should be performed to confirm active disease only if total HepBcAb is positive and HepBsAg is negative or if C antibody is positive,
* Myocardial infarction, stroke, transient ischemic attack (TIA), unstable angina, or coronary artery bypass surgery or other revascularization procedure within 12 months prior to screening,
* History or evidence of any other unstable or clinically significant medical condition that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion,
* Subject has any clinically significant vital sign, laboratory, or electrocardiogram (ECG) abnormality during screening that, in the opinion of the investigator, could pose a risk to subject safety or interfere with the study evaluation,
* The subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior or endorsing items 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) assessed at screening,
* Evidence of drug or alcohol abuse or dependence within 12 months prior to screening, based on medical records, patient self-report, or positive urine drug test performed during screening (with the exception of prescribed medications such as opioids or barbiturates),
* Pregnant or breastfeeding, or is a female expecting to conceive during the study, including through 16 weeks after the last dose of investigational product,
* Female subject of childbearing potential who is unwilling to use an acceptable method of effective contraception during treatment with investigational product through 16 weeks after the last dose of investigational product,
* Currently receiving treatment in another investigational device or drug study, or less than 90 days prior to screening since ending treatment on another investigational device or drug study(-ies),
* Known sensitivity to any component of the investigational product (Refer to the Investigational Product Instruction Manual [IPIM] for details),
* Previously randomized into an erenumab study,
* Member of investigational site staff or relative of the investigator,
* Unlikely to be able to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, independent completion of eDiary items) to the best of the subject's and investigator's knowledge.

Exclusion Criteria for the CHU Substudy:

- Unreliability as a study participant based on the investigator's (or designee's) knowledge of the subject (eg, unwillingness to adhere to the protocol, unwilling to self-inject using an autoinjector (AI)/pen after review of the Instructions for Use). Subjects receiving erenumab 70 mg in the open-label phase are not eligible.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (35):
- Japan (35):
  - Research Site, Kamogawa-shi, Chiba
  - Research Site, Saijo-shi, Ehime
  - Research Site, Ota-shi, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Kahoku-gun, Ishikawa-ken
  - Research Site, Morioka, Iwate
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Osaka, Osaka
  - Research Site, Osakasayama-shi, Osaka
  - Research Site, Toyonaka-shi, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Iruma-gun, Saitama
  - Research Site, Saitama-shi, Saitama
  - Research Site, Tokorozawa-shi, Saitama
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Shimotsuga-gun, Tochigi
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Chofu-shi, Tokyo
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Hachioji-shi, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Shibuya-ku, Tokyo
  - Research Site, Shinjuku-ku, Tokyo
  - Research Site, Yonago, Tottori
  - Research Site, Toyama, Toyama
  - Research Site, Hofu-shi, Yamaguchi
  - Research Site, Yamaguchi, Yamaguchi
  - Research Site, Kai-shi, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Sakai F, Takeshima T, Tatsuoka Y, Hirata K, Lenz R, Wang Y, Cheng S, Hirama T, Mikol DD. A Randomized Phase 2 Study of Erenumab for the Prevention of Episodic Migraine in Japanese Adults. Headache. 2019 Nov;59(10):1731-1742. doi: 10.1111/head.13652. Epub 2019 Oct 14. PMID 31612482
- [Background] Zhou Y, Zhang F, Starcevic Manning M, Hu Z, Hsu CP, Chen PW, Peng C, Loop B, Mytych DT, Paiva da Silva Lima G. Immunogenicity of erenumab: A pooled analysis of six placebo-controlled trials with long-term extensions. Cephalalgia. 2022 Jul;42(8):749-760. doi: 10.1177/03331024221075621. Epub 2022 Mar 10. PMID 35272533
- [Background] Hiramatsu K, Onizuka Y, Hasebe M, Yoshida R, Numachi Y. Novel Drug for Migraine Prophylaxis: Mode of Action, Efficacy and Safety of Erenumab. Shinryo to Shinyaku (Med Cons New-Remed) 2021:58(11):797-832
- [Background] Sakai F, Takeshima T, Tatsuoka Y, Hirata K, Cheng S, Numachi Y, Peng C, Xue F, Mikol DD. Long-term efficacy and safety during open-label erenumab treatment in Japanese patients with episodic migraine. Headache. 2021 Apr;61(4):653-661. doi: 10.1111/head.14096. Epub 2021 Mar 25. PMID 33764538
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study, initiated on 06 January 2016 at 43 centers in Japan, included a 24-week double-blind treatment phase (DBTP) followed by a 76-week open-label (OL) treatment phase (OLTP).
  DBTP: participants were randomized 2:1:2:2 to receive placebo, erenumab 28 mg, erenumab 70 mg, or erenumab 140 mg once monthly (QM) subcutaneously (SC).
Pre-assignment Details: OLTP: participants received erenumab 70 mg and/or 140 mg QM SC (depending on the participant's visit completion status after a protocol amendment).
  Optional 85-day clinical home use (CHU) sub-study during the OLTP: participants randomized 1:1 to erenumab using two 70 mg/mL or one 140 mg/mL autoinjector (AI)/pen(s).
Groups:
- DBTP: Placebo: Placebo SC on day 1 and at weeks 4, 8, 12, 16, and 20 in the DBTP.
- DBTP: Erenumab 28 mg QM: Erenumab 28 mg SC on day 1 and at weeks 4, 8, 12, 16, and 20 in the DBTP.
- DPTP: Erenumab 70 mg QM: Erenumab 70 mg SC on day 1 and at weeks 4, 8, 12, 16, and 20 in the DBTP.
- DBTP: Erenumab 140 mg QM: Erenumab 140 mg SC on day 1 and at weeks 4, 8, 12, 16, and 20 in the DBTP.
- OLTP: Erenumab 70 mg QM (Initial OL Dose): Participants assigned to an initial erenumab dose of 70 mg QM SC in the OLTP.
  After a protocol amendment, participants who had already completed the week 48 OLTP visit continued to receive OL erenumab 70 mg QM SC for a total of 76 weeks. Participants who had not yet completed the OLTP week 48 visit and were already receiving OL erenumab 70 mg QM SC increased their dose to erenumab 140 mg QM SC, continued until the week 100 visit for a total OLTP duration of 76 weeks.
- OLTP: Erenumab 140 mg QM (Initial OL Dose): Participants assigned to an initial erenumab dose of 140 mg QM SC in the OLTP.
  After a protocol amendment, participants who had not yet completed the DBTP and were not yet in the OLTP received an initial dose of erenumab 140 mg QM SC upon entering the OLTP, and continued receiving OL erenumab 140 mg QM SC for 76 weeks.
- CHU Sub-Study: Two 70 mg/mL AI/Pens: A subset of participants in the OLTP randomized to self-administer erenumab via two 70 mg/mL AI/pens on CHU sub-study day 1, day 29 and day 57.
- CHU Sub-Study: One 140 mg/mL AI/Pen: A subset of participants in the OLTP randomized to self-administer erenumab via one 140 mg/mL AI/pen on CHU sub-study day 1, day 29 and day 57.
Period: Double-Blind Treatment Phase (DBTP)
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM | OLTP: Erenumab 70 mg QM (Initial OL Dose) | OLTP: Erenumab 140 mg QM (Initial OL Dose) | CHU Sub-Study: Two 70 mg/mL AI/Pens | CHU Sub-Study: One 140 mg/mL AI/Pen
Started | 136 | 67 | 135 | 137 | 0 | 0 | 0 | 0
Received Investigational Product (IP) | 136 | 66 | 135 | 137 | 0 | 0 | 0 | 0
Completed (Completed week 24 assessment of double-blind treatment phase) | 133 | 65 | 130 | 134 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 5 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol-specified criteria | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Sponsor decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 4 | 1 | 0 | 0 | 0 | 0
Not completed — Subject missed week 24 assessment | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-Label Treatment Phase (OLTP)
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM | OLTP: Erenumab 70 mg QM (Initial OL Dose) | OLTP: Erenumab 140 mg QM (Initial OL Dose) | CHU Sub-Study: Two 70 mg/mL AI/Pens | CHU Sub-Study: One 140 mg/mL AI/Pen
Started | 0 | 0 | 0 | 0 | 386 | 73 | 0 | 0
Received Only 70 mg in OLTP | 0 | 0 | 0 | 0 | 270 | 0 | 0 | 0
Received Only 140 mg in OLTP | 0 | 0 | 0 | 0 | 0 | 73 | 0 | 0
Received Both 70 mg and 140 mg in OLTP | 0 | 0 | 0 | 0 | 116 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 357 | 69 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 29 | 4 | 0 | 0
Not completed — Protocol-Specified Criteria | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0
Not completed — Subject Request | 0 | 0 | 0 | 0 | 24 | 3 | 0 | 0
Not completed — Decision by Sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Optional CHU Sub-Study (During OLTP)
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM | OLTP: Erenumab 70 mg QM (Initial OL Dose) | OLTP: Erenumab 140 mg QM (Initial OL Dose) | CHU Sub-Study: Two 70 mg/mL AI/Pens | CHU Sub-Study: One 140 mg/mL AI/Pen
Started | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 25
Completed (Completed week 12 sub-study visit (day 85)) | 0 | 0 | 0 | 0 | 0 | 0 | 24 | 25
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM | Total
Number analyzed (Participants) | 136 | 67 | 135 | 137 | 475
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.7 (9.1) | 42.8 (6.9) | 43.8 (9.0) | 45.0 (8.3) | 44.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 55 | 115 | 112 | 400
  Male | 18 | 12 | 20 | 25 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 136 | 67 | 135 | 137 | 475
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 136 | 67 | 135 | 137 | 475
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Monthly Migraine Days at Baseline [Mean (Standard Deviation); unit: Days] — The number of migraine days in the 4-week baseline period. A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation or recurrence of the migraine headache). A qualified migraine headache was defined as a migraine with or without aura, lasting for ≥ 30 minutes and meeting at least one of the pre-specified pain features and/or associated symptoms criteria.
  Days | 7.67 (2.34) | 7.68 (2.14) | 7.84 (2.31) | 8.14 (2.43) | 7.86 (2.33)
Treatment Status with Migraine Prophylactic Medication [Count of Participants; unit: Participants] — Treatment status values presented are those utilized in the randomization process.
  Participants
    Current treatment | 14 | 7 | 13 | 15 | 49
    Prior treatment only | 75 | 38 | 75 | 75 | 263
    No prior or current treatment | 47 | 22 | 47 | 47 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Monthly Migraine Days at Months 4, 5 and 6
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation or recurrence of the migraine headache). A qualified migraine headache was a migraine with or without aura, lasting for ≥ 30 minutes, and meeting at least one of the following criteria: a) ≥ 2 of the following pain features: unilateral, throbbing, moderate to severe, exacerbated with exercise/physical activity; b) ≥ 1 of the following associated symptoms: nausea and/or vomiting, photophobia and phonophobia. Change from baseline was calculated using the mean monthly migraine days from months 4, 5 and 6 of the DBTP minus the number of migraine days during the 4-week baseline phase. Least squares (LS) mean was estimated using a generalized linear mixed model which included treatment, visit, treatment by visit interaction, stratification factor (current, prior only, or no prior/current treatment), and baseline value as covariates.
Time Frame: 4-week baseline phase and months 4, 5 and 6 of DBTP.
Population: Efficacy Analysis Set: Participants who received at least 1 dose of the investigational product (IP) and had at least 1 change from baseline measurement in monthly migraine days during the DBTP.
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM
Number analyzed (Participants) | 136 | 66 | 135 | 136
Days | 0.06 [-0.46 to 0.58] | -1.19 [-1.91 to -0.47] | -2.25 [-2.78 to -1.73] | -1.83 [-2.35 to -1.31]
Statistical Analysis 1: Comparison: DBTP: Placebo vs DBTP: Erenumab 140 mg QM; The primary analysis utilized a generalized linear mixed model which included treatment, visit, treatment by visit interaction, stratification factor (prior/current treatment with migraine prophylactic medication status), and baseline value as covariates and assumed a first-order autoregressive covariance structure; Test type: Superiority — To maintain a family-wise type I error at 0.05, the pairwise comparisons were tested in a sequential testing procedure in the order of erenumab 140 mg QM vs placebo, erenumab 70 mg QM vs placebo and erenumab 28 mg QM vs placebo. The lower dose group was tested only when the higher dose group was considered statistically significant; p < 0.001, Generalized Linear Mixed Model — P-values for pairwise comparisons were nominal and without multiplicity adjustment; LS Mean Difference = -1.89, 95% CI 2-sided [-2.58 to -1.20]
Statistical Analysis 2: Comparison: DBTP: Placebo vs DPTP: Erenumab 70 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Generalized Linear Mixed Model — P-values for pairwise comparisons were nominal and without multiplicity adjustment; LS Mean Difference = -2.31, 95% CI 2-sided [-3.00 to -1.62]
Statistical Analysis 3: Comparison: DBTP: Placebo vs DBTP: Erenumab 28 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.004, Generalized Linear Mixed Model — P-values for pairwise comparisons were nominal and without multiplicity adjustment; LS Mean Difference = -1.25, 95% CI 2-sided [-2.10 to -0.41]

2. Primary Outcome: CHU Sub-Study: Participant-Reported Outcome of Attempted Full-Dose Administration at Day 29 (Week 4) and Day 57 (Week 8)
Description: On CHU day 29 and day 57, site staff interviewed sub-study participants and asked if they administered a full, partial, or no dose of erenumab (after explaining that a full dose means that the entire volume of the AI/pen was injected) and documented the participant's response in the electronic case report form. Data presented are the percentage of participants who reported "full administration," "not full administration," or "discontinued investigational product (ie, no dose)." (Day 1 of the CHU substudy occurred at any OLTP study visit [up to week 88] as long as the participant had previously received at least 1 OL dose of erenumab 140 mg.)
Time Frame: CHU day 29 (week 4) and day 57 (week 8)
Population: CHU Sub-Study Analysis Set: all participants randomized into the CHU substudy who received at least one dose of CHU investigational product (IP).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CHU Sub-Study: Two 70 mg/mL AI/Pens | CHU Sub-Study: One 140 mg/mL AI/Pen
Number analyzed (Participants) | 24 | 25
percentage of participants
  Week 4: Full Administration | 100.0 [86.2 to 100.0] | 100.0 [86.7 to 100.0]
  Week 4: Not Full Administration | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 13.3]
  Week 4: Discontinued Investigational Product | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 13.3]
  Week 8: Full Administration | 100.0 [86.2 to 100.0] | 100.0 [86.7 to 100.0]
  Week 8: Not Full Administration | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 13.3]
  Week 8: Discontinued Investigational Product | 0.0 [0.0 to 13.8] | 0.0 [0.0 to 13.3]
Statistical Analysis 1: Comparison: CHU Sub-Study: Two 70 mg/mL AI/Pens vs CHU Sub-Study: One 140 mg/mL AI/Pen; Week 4: Full Administration; Test type: Superiority; Treatment Difference = 0.0, 95% CI 2-sided [-13.3 to 13.8] — The 95% CI for the difference was calculated using the Newcombe hybrid score method
Statistical Analysis 2: Comparison: CHU Sub-Study: Two 70 mg/mL AI/Pens vs CHU Sub-Study: One 140 mg/mL AI/Pen; Week 4: Not Full Administration; Test type: Superiority; Treatment Difference = 0.0, 95% CI 2-sided [-13.8 to 13.3] — The 95% CI for the difference was calculated using the Newcombe hybrid score method
Statistical Analysis 3: Comparison: CHU Sub-Study: Two 70 mg/mL AI/Pens vs CHU Sub-Study: One 140 mg/mL AI/Pen; Week 4: Discontinued Investigational Product; Test type: Superiority; Treatment Difference = 0.0, 95% CI 2-sided [-13.8 to 13.3] — The 95% CI for the difference was calculated using the Newcombe hybrid score method
Statistical Analysis 4: Comparison: CHU Sub-Study: Two 70 mg/mL AI/Pens vs CHU Sub-Study: One 140 mg/mL AI/Pen; Week 8: Full Administration; Test type: Superiority; Treatment Difference = 0.0, 95% CI 2-sided [-13.3 to 13.8] — The 95% CI for the difference was calculated using the Newcombe hybrid score method
Statistical Analysis 5: Comparison: CHU Sub-Study: Two 70 mg/mL AI/Pens vs CHU Sub-Study: One 140 mg/mL AI/Pen; Week 8: Not Full Administration; Test type: Superiority; Treatment Difference = 0.0, 95% CI 2-sided [-13.8 to 13.3] — The 95% CI for the difference was calculated using the Newcombe hybrid score method
Statistical Analysis 6: Comparison: CHU Sub-Study: Two 70 mg/mL AI/Pens vs CHU Sub-Study: One 140 mg/mL AI/Pen; Week 8: Discontinued Investigational Product; Test type: Superiority; Treatment Difference = 0.0, 95% CI 2-sided [-13.8 to 13.3] — The 95% CI for the difference was calculated using the Newcombe hybrid score method

3. Secondary Outcome: Percentage of Participants With at Least a 50% Reduction From Baseline in Mean Monthly Migraine Days at Months 4, 5 and 6
Description: A migraine day was defined as any calendar day in which the participant experienced a qualified migraine headache (onset, continuation or recurrence of the migraine headache). A qualified migraine headache was a migraine with or without aura, lasting for ≥ 30 minutes, and meeting at least one of the following criteria: a) ≥ 2 of the following pain features: unilateral, throbbing, moderate to severe, exacerbated with exercise/physical activity; b) ≥ 1 of the following associated symptoms: nausea and/or vomiting, photophobia and phonophobia.
  At least a 50% reduction from baseline in monthly migraine days was determined if: (mean monthly migraine days over the last three months of the DBTP minus baseline monthly migraine days) * 100 / baseline monthly migraine days, was less than or equal to -50%.
Time Frame: 4-week baseline phase and months 4, 5 and 6 of DBTP.
Population: Efficacy Analysis Set: Participants who received at least 1 dose of IP and had at least 1 change from baseline measurement in monthly migraine days during the DBTP.
Measure: Number; unit: Percentage of participants
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM
Number analyzed (Participants) | 136 | 66 | 135 | 136
Percentage of participants | 7.4 | 19.7 | 28.9 | 27.2
Statistical Analysis 1: Comparison: DBTP: Placebo vs DBTP: Erenumab 140 mg QM; The common odds ratios and p-values were obtained from a Cochran-Mantel-Haenszel (CMH) test, stratified by stratification factor prior/current treatment with migraine prophylactic medication status; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for pairwise comparisons were nominal and obtained from the CMH test using data including placebo and corresponding erenumab dose group only; Common Odds Ratio = 4.73, 95% CI 2-sided [2.24 to 9.99]
Statistical Analysis 2: Comparison: DBTP: Placebo vs DPTP: Erenumab 70 mg QM; The common odds ratios and p-values were obtained from a CMH test, stratified by stratification factor prior/current treatment with migraine prophylactic medication status; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Common Odds Ratio = 5.60, 95% CI 2-sided [2.60 to 12.06]
Statistical Analysis 3: Comparison: DBTP: Placebo vs DBTP: Erenumab 28 mg QM; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Common Odds Ratio = 3.21, 95% CI 2-sided [1.30 to 7.88]

4. Secondary Outcome: Change From Baseline in Mean Monthly Acute Migraine-Specific Medication Treatment Days at Months 4, 5 and 6
Description: An acute migraine-specific medication treatment day was defined as any calendar day during which the participant took a migraine-specific medication (ie, triptan or ergotamine-derivatives).
  The change from baseline was calculated using the mean monthly acute migraine-specific medication treatment days over the last three months (months 4, 5 and 6) of the DBTP minus the baseline monthly acute migraine-specific medication treatment days.
  LS mean was estimated using a generalized linear mixed model which included treatment, visit, treatment by visit interaction, stratification factor (prior/current treatment), and baseline value as covariates.
Time Frame: 4-week baseline phase and months 4, 5 and 6 of DBTP.
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM
Number analyzed (Participants) | 136 | 66 | 135 | 136
Days | 0.88 [0.44 to 1.33] | -0.19 [-0.80 to 0.43] | -1.19 [-1.64 to -0.74] | -1.16 [-1.60 to -0.71]
Statistical Analysis 1: Comparison: DBTP: Placebo vs DBTP: Erenumab 140 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Generalized Linear Mixed Model — P-values for pairwise comparisons were nominal and without multiplicity adjustment; LS Mean Difference = -2.04, 95% CI 2-sided [-2.63 to -1.45]
Statistical Analysis 2: Comparison: DBTP: Placebo vs DPTP: Erenumab 70 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Generalized Linear Mixed Model — P-values for pairwise comparisons were nominal and without multiplicity adjustment; LS Mean Difference = -2.07, 95% CI 2-sided [-2.66 to -1.49]
Statistical Analysis 3: Comparison: DBTP: Placebo vs DBTP: Erenumab 28 mg QM; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.004, Generalized Linear Mixed Model — P-values for pairwise comparisons were nominal and without multiplicity adjustment; LS Mean Difference = -1.07, 95% CI 2-sided [-1.80 to -0.35]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Discontinuations Due to TEAEs, and Fatal TEAEs During the DBTP
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. A serious adverse event (SAE) is defined as an adverse event that meets at least 1 of the following serious criteria: fatal; life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious event. Events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 (grade 1=mild, grade 2=moderate, grade 3=severe, grade 4= life-threatening, grade 5=death).
Time Frame: From first dose of IP up to week 24
Population: Safety Analysis Set: all randomized participants who received at least one dose of IP in the DBTP.
Measure: Count of Participants; unit: Participants
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM
Number analyzed (Participants) | 136 | 66 | 135 | 137
Participants
  All TEAEs | 92 | 40 | 95 | 95
  Grade ≥ 2 TEAEs | 60 | 33 | 66 | 65
  Grade ≥ 3 TEAEs | 4 | 1 | 3 | 0
  Grade ≥ 4 TEAEs | 0 | 0 | 1 | 0
  Serious TEAEs | 4 | 1 | 1 | 1
  TEAEs Leading to Discontinuation of IP | 1 | 0 | 2 | 0
  Fatal TEAEs | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs, Discontinuations Due to TEAEs, and Fatal TEAEs During the OLTP
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant. An SAE is defined as an adverse event that meets at least 1 of the following serious criteria: fatal; life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious event. Events were graded according to the NCI CTCAE version 4.03 (grade 1=mild, grade 2=moderate, grade 3=severe, grade 4= life-threatening, grade 5=death).
Time Frame: From first dose of IP in the OLTP (week 24) through the end of the OLTP (week 100) plus 12 weeks
Population: Open-Label Treatment Phase Set: all participants receiving at least one dose of IP in the OLTP, by dose received at the time of the event, and overall (total participants in the OLTP).
Measure: Count of Participants; unit: Participants
Groups:
- OLTP: Erenumab 70 mg QM: Erenumab 70 mg SC QM in the OLTP (at the time of the event).
- OLTP: Erenumab 140 mg QM: Erenumab 140 mg SC QM in the OLTP (at the time of the event).
- OLTP: Total: Participants receiving erenumab 70 mg and/or 140 mg SC QM in the OLTP
Arm/Group | OLTP: Erenumab 70 mg QM | OLTP: Erenumab 140 mg QM | OLTP: Total
Number analyzed (Participants) | 386 | 189 | 459
Participants
  All TEAEs | 292 | 173 | 422
  Grade ≥ 2 TEAEs | 238 | 147 | 358
  Grade ≥ 3 TEAEs | 19 | 9 | 28
  Grade ≥ 4 TEAEs | 0 | 0 | 0
  Serious TEAEs | 18 | 9 | 27
  TEAEs Leading to Discontinuation of IP | 4 | 2 | 6
  Fatal TEAEs | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs, Discotninuations Due to TEAEs, Fatal TEAEs, and Adverse Device Effects During the CHU Sub-Study
Description: An AE is defined as any untoward medical occurrence in a clinical trial participant. An SAE is defined as an adverse event that meets at least 1 of the following serious criteria: fatal; life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; congenital anomaly/birth defect; other medically important serious event. Events were graded according to the NCI CTCAE version 4.03 (grade 1=mild, grade 2=moderate, grade 3=severe, grade 4= life-threatening, grade 5=death). TEAEs leading to discontinuation of IP are TEAEs leading to complete discontinuation of erenumab regardless of CHU IP or parent study IP.
Time Frame: CHU sub-study day 1 through day 85 (end of CHU sub-study). Day 1 of the CHU substudy occurred at any OLTP study visit (up to week 88) as long as the participant had previously received at least 1 OL dose of erenumab 140 mg.
Population: CHU Sub-Study Analysis Set: all participants randomized into the CHU substudy who received at least one dose of CHU IP.
Measure: Count of Participants; unit: Participants
Arm/Group | CHU Sub-Study: Two 70 mg/mL AI/Pens | CHU Sub-Study: One 140 mg/mL AI/Pen
Number analyzed (Participants) | 24 | 25
Participants
  All TEAEs | 11 | 14
  Grade ≥ 2 TEAEs | 9 | 9
  Grade ≥ 3 TEAEs | 0 | 0
  Grade ≥ 4 TEAEs | 0 | 0
  Serious TEAEs | 1 | 0
  TEAEs Leading to Discontinuation of IP | 0 | 0
  Fatal TEAEs | 0 | 0
  Adverse Device Effects | 2 | 1

8. Secondary Outcome: Number of Participants With Post-Baseline Liver Function Test Abnormalities During the DBTP
Description: Post-baseline is defined as any assessment done after the first dose of IP. Liver Function tests included alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin (TBL). ULN=upper limit of normal.
Time Frame: From the first dose of study IP through the end of the DBTP (up to week 24)
Population: Safety Analysis Set: all randomized participants who received at least one dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM
Number analyzed (Participants) | 136 | 66 | 135 | 137
Participants
  Post-Baseline ALT or AST > 3 x ULN | 0 | 0 | 3 | 1
  Post-Baseline ALT or AST > 5 x ULN | 0 | 0 | 0 | 1
  Post-Baseline TBL > 1 x ULN | 6 | 3 | 4 | 4
  Post-Baseline TBL > 1.5 x ULN | 0 | 1 | 0 | 1
  Post-Baseline TBL > 2 x ULN | 0 | 0 | 0 | 0
  Post-Baseline ALP > 1.5 x ULN | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Post-Baseline Liver Function Test Abnormalities During the OLTP
Description: Post-baseline is defined as any assessment done after the first dose of OLTP IP. Liver Function tests included alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin (TBL). ULN=upper limit of normal.
Time Frame: From the first dose of OLTP IP (week 24) through the end of the OLTP (up to week 100)
Population: Safety Analysis Set: all randomized participants who received at least one dose of OLTP erenumab.
Measure: Count of Participants; unit: Participants
Groups:
- OLTP: 70 mg SC QM (Only): Participants who received only erenumab 70 mg SC QM in the OLTP
- OLTP: 140 mg SC QM (Only): Participants who received only erenumab 140 mg SC QM in the OLTP
- OLTP: 70/140 mg SC QM (Both): Participants who received both erenumab 70 mg and 140 mg SC QM in the OLTP
- OLTP: Total: Participants who received erenumab 70 mg and/or 140 mg SC QM in the OLTP
Arm/Group | OLTP: 70 mg SC QM (Only) | OLTP: 140 mg SC QM (Only) | OLTP: 70/140 mg SC QM (Both) | OLTP: Total
Number analyzed (Participants) | 270 | 73 | 116 | 459
Participants
  Post-Baseline ALT or AST > 3 x ULN | 4 | 2 | 0 | 6
  Post-Baseline ALT or AST > 5 x ULN | 0 | 0 | 0 | 0
  Post-Baseline TBL > 1 x ULN | 12 | 3 | 6 | 21
  Post-Baseline TBL > 1.5 x ULN | 0 | 0 | 0 | 0
  Post-Baseline TBL > 2 x ULN | 0 | 0 | 0 | 0
  Post-Baseline ALP > 1.5 x ULN | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Blood Pressure Changes From Baseline in Categories at Week 24 During the DBTP
Description: Participants with increases (↑) from baseline (BL) in diastolic blood pressure (DBP) and systolic blood pressure (SBP) at week 24 (Wk24) are presented.
Time Frame: Baseline (last assessment prior to first dose of IP), week 24
Population: Safety Analysis Set: all randomized participants who received at least one dose of IP. Participants with an assessment at week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM
Number analyzed (Participants) | 135 | 65 | 130 | 134
Participants
  ↑ from BL ≥10 mmHg in DBP w/DBP >90 mmHg at Wk24 | 3 | 2 | 1 | 3
  ↑ from BL ≥10 mmHg in DBP w/DBP ≤90 mmHg at Wk24 | 14 | 6 | 14 | 8
  ↑ from BL ≥20 mmHg in SBP w/SBP >140 mmHg at Wk24 | 1 | 1 | 0 | 2
  ↑ from BL ≥20 mmHg in SBP w/SBP ≤140 mmHg at Wk24 | 0 | 2 | 0 | 3

11. Secondary Outcome: Number of Participants With Blood Pressure Changes From Pre-OLTP Baseline in Categories at Week 100 During the OLTP
Description: Participants with increases (↑) from baseline (BL) in diastolic blood pressure (DBP) and systolic blood pressure (SBP) at week 100 (Wk100) are presented.
Time Frame: Pre-OLTP Baseline (last assessment prior to first dose of IP in OLTP), week 100
Population: Safety Analysis Set: all randomized participants who received at least one dose of IP in the OLTP. Participants with an assessment at week 100.
Measure: Count of Participants; unit: Participants
Arm/Group | OLTP: 70 mg SC QM (Only) | OLTP: 140 mg SC QM (Only) | OLTP: 70/140 mg SC QM (Both) | OLTP: Total
Number analyzed (Participants) | 245 | 68 | 112 | 425
Participants
  ↑ from BL ≥10 mmHg in DBP w/DBP >90 mmHg at Wk100 | 8 | 0 | 2 | 10
  ↑ from BL ≥10 mmHg in DBP w/DBP ≤90 mmHg at Wk100 | 25 | 10 | 10 | 45
  ↑ from BL ≥20 mmHg in SBP w/SBP >140 mmHg at Wk100 | 4 | 0 | 1 | 5
  ↑ from BL ≥20 mmHg in SBP w/SBP ≤140 mmHg at Wk100 | 7 | 2 | 0 | 9

12. Secondary Outcome: Number of Participants With Anti-Erenumab Antibodies During the Entire Study for Participants Who Received ≥ 1 Dose of Erenumab
Description: Data are summarized by the treatment participants received during the double-blind treatment phase. Placebo participants may have received erenumab 70 mg or 140 mg during the OLTP. Baseline is defined as the last antibody assessment on or prior to the first dose of erenumab.
  Transient binding/neutralizing antibody responses are defined as a negative (neg) result at the participant's last timepoint tested among participants who developed binding/neutralizing antibodies post-baseline.
Time Frame: Baseline (first dose of erenumab) up to end of study (week 100) plus 12 weeks
Population: Safety Analysis Set: all randomized participants who received at least one dose of IP. Participants who received at least one dose of erenumab (during the DBTP and/or OLTP).
Measure: Count of Participants; unit: Participants
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM
Number analyzed (Participants) | 133 | 66 | 135 | 137
Participants
  Binding Antibody Positive (BAb+) at Baseline (BL) | 0 | 0 | 0 | 0
  Neutralizing Antibody Positive (NAb+) at BL | 0 | 0 | 0 | 0
  BAb+ Post-BL With a Neg/No Result at BL | 4 | 5 | 6 | 0
  Transient BAb+ Post-BL With a Neg/No Result at BL | 2 | 4 | 5 | 0
  NAb+ Post-BL With a Neg/No Result at BL | 0 | 0 | 0 | 0
  Transient NAb+ Post-BL With a Neg/No Result at BL | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: from randomization through the end of study (up to 116 weeks). Treatment-emergent serious and non-serious events: - DBTP: from first dose of IP up to week 24 (end of DBTP) - OLTP: from first dose of OL IP (week 24) up to week 100 (end of OLTP) plus 12 weeks - CHU sub-study: from first dose of sub-study IP up to day 85 (end of sub-study)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- OLTP Total: Erenumab 70/140 mg QM: Erenumab 70 mg and/or 140 mg SC QM in the OLTP.
- CHU Sub-Study: Two Erenumab 70 mg/mL AI/Pens: Self-administered erenumab via two 70 mg/mL AI/pens on day 1, day 29 and day 57 of the CHU sub-study.
- CHU Sub-Study: One Erenumab 140 mg/mL AI/Pen: Self-administered erenumab via one 140 mg/mL AI/pen on day 1, day 29 and day 57 of the CHU sub-study.
- CHU Sub-Study Total: Self-administered erenumab via two 70 mg/mL AI/pens or one 140 mg/mL AI/pen on day 1, day 29 and day 57 of the CHU sub-study.
Arm/Group | DBTP: Placebo | DBTP: Erenumab 28 mg QM | DPTP: Erenumab 70 mg QM | DBTP: Erenumab 140 mg QM | OLTP: Erenumab 70 mg QM | OLTP: Erenumab 140 mg QM | OLTP Total: Erenumab 70/140 mg QM | CHU Sub-Study: Two Erenumab 70 mg/mL AI/Pens | CHU Sub-Study: One Erenumab 140 mg/mL AI/Pen | CHU Sub-Study Total
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/67 | 0/135 | 0/137 | 0/386 | 0/189 | 0/459 | 0/24 | 0/25 | 0/49
Serious Adverse Events (participants affected / at risk) | 4/136 | 1/66 | 1/135 | 1/137 | 18/386 | 9/189 | 27/459 | 1/24 | 0/25 | 1/49
Other Adverse Events (participants affected / at risk) | 55/136 | 28/66 | 67/135 | 58/137 | 231/386 | 133/189 | 343/459 | 7/24 | 7/25 | 14/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DBTP: Placebo (N=136) | DBTP: Erenumab 28 mg QM (N=66) | DPTP: Erenumab 70 mg QM (N=135) | DBTP: Erenumab 140 mg QM (N=137) | OLTP: Erenumab 70 mg QM (N=386) | OLTP: Erenumab 140 mg QM (N=189) | OLTP Total: Erenumab 70/140 mg QM (N=459) | CHU Sub-Study: Two Erenumab 70 mg/mL AI/Pens (N=24) | CHU Sub-Study: One Erenumab 140 mg/mL AI/Pen (N=25) | CHU Sub-Study Total (N=49)
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Extremity contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Myelopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBTP: Placebo (N=136) | DBTP: Erenumab 28 mg QM (N=66) | DPTP: Erenumab 70 mg QM (N=135) | DBTP: Erenumab 140 mg QM (N=137) | OLTP: Erenumab 70 mg QM (N=386) | OLTP: Erenumab 140 mg QM (N=189) | OLTP Total: Erenumab 70/140 mg QM (N=459) | CHU Sub-Study: Two Erenumab 70 mg/mL AI/Pens (N=24) | CHU Sub-Study: One Erenumab 140 mg/mL AI/Pen (N=25) | CHU Sub-Study Total (N=49)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 5 | 2 | 22 | 4 | 26 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 7 | 7 | 14 | 5 | 19 | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 3 | 2 | 7 | 2 | 17 | 9 | 26 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 2 | 2 | 4 | 27 | 15 | 41 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 41 | 22 | 39 | 45 | 174 | 109 | 274 | 5 | 6 | 11
Pharyngitis (Infections and infestations) | 3 | 3 | 5 | 3 | 22 | 7 | 28 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 7 | 1 | 28 | 7 | 34 | 1 | 0 | 1
Cystitis (Infections and infestations) | 3 | 1 | 1 | 2 | 18 | 8 | 26 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 1 | 3 | 1 | 46 | 29 | 75 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02630459/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT02630459/SAP_001.pdf